CLINICAL TRIAL: NCT01834417
Title: Preliminary Study Leading to Prevention of Pressure Ulcers by the Use of an On-board Device : Ergonomic Assessment of Wheelchair-seat Pressures in Spinal Cord Injured (SCI) Patients
Brief Title: Preliminary Study Leading to Prevention of Pressure Ulcers by the Use of an On-board Device : Ergonomic Assessment of Wheelchair-seat Pressures in Spinal Cord Injured (SCI) Patients ( PRESDIE)
Acronym: PRESDIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC11_0009
Record Dates: First submitted 2013-04-08; First posted 2013-04-17 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Pressure Ulcer
Keywords: Pressure ulcer, spinal cord injury, on-board device
MeSH Terms: conditions — Pressure Ulcer; Spinal Cord Injuries

INTERVENTIONS:
Device: TexiMat

SUMMARY:
Analysis of stored seat-pressures in SCI patients during a 4-week use of an on-board device. During this period, patients write in an agenda noteworthy events that could occur while they're using their wheelchair. A control is done every week and the device can be changed until it is returned at the end of the study period.

DETAILED DESCRIPTION:
* inclusion visit : recovery of the signed informed-consent form, clinical examination, skin control, seat-pressures control, device 9-position control, delivery of the agenda for noteworthy events
* 3 follow-up visits : noteworthy events check, skin control, cushioncloth control, device 9-position control
* return visit : device return, agenda return, skin control, seat-pressures control

ELIGIBILITY:
Inclusion criteria :

* Patient is male or female, aged ≥ 18
* Patient accepting the initial assessment and the following visits during the protocol
* Written informed consent has been obtained
* Patient having a social assurance
* Spinal cord injury ≤ C6 stable Spinal cord trauma > 1 an
* Main mode of ambulation : own manual wheelchair

Exclusion criteria :

* Aged ≤ 18
* Adults under guardianship
* Patients do not speak French, refusing or unable to be followed
* Pregnant or lactating women
* Person deprived of their liberty by judicial or administrative decision
* Person hospitalised without consent
* Pelvic pressure ulcer ongoing
* Cognitive disorder incompatible with the use of the device, understanding and conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-04-18 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Intra- and inter-patients variability of stored pressures for the whole included population Intra- and inter-patients variability of stored pressures for the whole included population | 4 weeks
  Intra- and inter-patients variability of stored pressures for the whole included population Measured at the end of the study
  Each topic will be equipped with a layer of pressure sensors 32x32. The pressure maps are stored every second rule, which will be of the order of 30 000 maps daily. For each topic, we will be able to calculate the frequency and location of peak pressure

SECONDARY OUTCOMES:
Intra- and inter-patients variability of stored pressures for subpopulations | 4 weeks
  Intra- and inter-patients variability of stored pressures for subpopulations :
  * quadriplegic vs paraplegic
  * according to high-risk areas for pressure ulcers
  * according to noteworthy events
  Each topic will be equipped with a layer of pressure sensors 32x32. The pressure maps are stored every second rule, which will be of the order of 30 000 maps daily. For each topic, we will be able to calculate the frequency and location of peak pressure Measured at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte PERROUIN-VERBE, PU-PH, Principal Investigator — CHU de Nantes- Hôpital Saint Jacques; Marc Le Fort, PH, Study Chair — CHU de Nantes-Hôpital Saint Jacques; Guy Egon, Study Chair — Centre de l'Arche; Djamel Bensmail, PU-PH, Study Chair — CH Raymond Poincaré
Locations (1):
- CHU Nantes, Nantes, France